CLINICAL TRIAL: NCT03926195
Title: A Randomized, Double-blind, Placebo-controlled Phase 2 Study to Evaluate the Effect of Filgotinib on Semen Parameters in Adult Males With Active Rheumatoid Arthritis, Psoriatic Arthritis, Ankylosing Spondylitis or Non-radiographic Axial Spondyloarthritis
Brief Title: Study to Evaluate the Effect of Filgotinib on Semen Parameters in Adult Males With Active Rheumatoid Arthritis, Psoriatic Arthritis, Ankylosing Spondylitis, or Non-radiographic Axial Spondyloarthritis
Acronym: MANTA-RAy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GLPG0634-CL-227; 2018-003933-14 (EudraCT Number)
Record Dates: First submitted 2019-04-19; First posted 2019-04-24 (Actual); Results first posted 2023-08-01 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Rheumatoid Arthritis; Psoriatic Arthritis; Ankylosing Spondylitis; Non-Radiographical Axial Spondyloarthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Psoriatic; Spondylitis, Ankylosing | interventions — GLPG0634; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Filgotinib (Experimental): Participants received filgotinib 200 milligrams (mg) tablet, orally, once daily up to Week 13 in the double-blind (DB) phase. At Week 13, participants who were arthritis responders, were unblinded and received open-label (OL) treatment filgotinib 200 mg, tablet, orally, once daily up to approximately 143 weeks (until Week 156) in the extension (EXT) phase and participants who were arthritis nonresponders discontinued blinded study drug and started standard of care (SOC) treatment in the EXT phase. Participants on DB treatment or OL filgotinib who entered the monitoring phase (if their sperm parameters met ≥50% decrease threshold in pre-specified semen parameters) discontinued the study drug and started SOC for up to 52 weeks.
  Interventions: Drug: Filgotinib; Drug: Standard of Care
- Placebo (Placebo Comparator): Participants received placebo (matched to filgotinib) tablet, orally, once daily up to Week 13 in the DB phase. At Week 13, participants were unblinded and started SOC treatment in the EXT phase for up to approximately 143 weeks (until Week 156). Participants who entered the monitoring phase (if their sperm parameters met ≥50% decrease threshold in pre-specified semen parameters) continued on SOC treatment.
  Interventions: Drug: Placebo; Drug: Standard of Care

INTERVENTIONS:
Drug: Filgotinib — 200-mg tablet administered orally once daily
  Other Names: GS-6034; Jyseleca®
  Arms: Filgotinib
Drug: Placebo — Placebo to match filgotinib tablet administered orally once daily
  Arms: Placebo
Drug: Standard of Care — Locally approved treatment, accepted by medical experts as a proper treatment for rheumatic conditions, prescribed according to best clinical practice, with no known testicular toxicity.

SUMMARY:
The primary objective of this study is to evaluate the effect of filgotinib on semen parameters in adult males with active rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, or non-radiographic axial spondyloarthritis.

Results of this study may be pooled with the results of a separate study being conducted in participants with inflammatory bowel disease (Protocol GS-US-418-4279; NCT03201445) with the same objective.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of active rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis or, non-radiographic axial spondyloarthritis for at least 12 weeks prior to screening, meeting the corresponding specific disease classification criteria as specified in the protocol

Key Exclusion Criteria:

* Previously documented problems with male reproductive health
* Prior diagnosis of male infertility
* Use of any prohibited concomitant medication as outlined by protocol

Note: Other protocol-defined Inclusion/Exclusion criteria may apply.

Ages: 21 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2019-05-28 (Actual); Primary Completion 2020-08-14 (Actual); Study Completion 2023-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Galapagos Study Director, Study Director — Galapagos NV
Locations (71):
- Bulgaria (12):
  - Medical center Medconsult Pleven OOD, Pleven
  - UMHAT Pulmed OOD, Plovdiv
  - UMHAT Sv. Georgi, EAD, Plovdiv
  - MHAT "Eurohospital" - Plovdiv, OOD, Plovdiv
  - Medical Center Teodora, EOOD, Rousse
  - Medizinski Zentar-1-Sevlievo EOOD, Sevlievo
  - Medical Center Excelsior, OOD, Sofia
  - DCC Alexandrovska, EOOD, Sofia
  - UMHAT Sv. Ivan Rilski, EAD, Sofia
  - DCC 17 - Sofia EOOD, Sofia
  - Meditsinski Centar - Izgrev EOOD, Sofia
  - MC Synexus - Sofia, EOOD, Sofia
- Czechia (11):
  - CCR Brno S.r.o., Brno
  - CCBR Ostrava s.r.o, Ostrava
  - Vesalion s.r.o., Ostrava
  - MUDr. Rosypalova s.r.o., Ostrava
  - Bioclinica Pardubice, Pardubice
  - CLINTRIAL s.r.o., Prague
  - Revmatologicky Ustav, Prague
  - Thomayerova nemocnice, Prague
  - MUDr Zuzana Stejfova Revmatologicka ambulance, Prague
  - Affidea Praha s.r.o., Prague
  - MEDICAL PLUS s.r.o., Uherské Hradiště
- Estonia (5):
  - OÜ Innomedica, Tallinn
  - Center for Clinical and Basic Research, Tallinn
  - North Estonia Medical Centre Foundation, Tallinn
  - Clinical Research Centre, Tartu
  - Meditrials OU, Tartu
- Georgia (8):
  - Chapidze Emergency Cardiology Center, Tbilisi
  - Institute of Clinical Cardiology Ltd, Tbilisi
  - National Institute of Endocrinology, Tbilisi
  - Tbilisi Heart and Vascular Clinic Ltd, Tbilisi
  - Aversi ClinicLtd., Tbilisi
  - Clinic on Mtskheta Street, Tbilisi
  - Consilium Medulla-multiprofile clinic Ltd, Tbilisi
  - Medicore Ltd., Tbilisi
- M&M center, Ādaži, Latvia
- Poland (12):
  - Nasz Lekarz Osrodek Badan Klinicznych, Bydgoszcz
  - Szpital Uniwersytecki nr 2 im. dr J. Biziela, Bydgoszcz
  - Silmedic sp. z o.o, Katowice
  - Indywidualna Specjalistyczna Praktyka Lekarska Maciej Zymla, Knurów
  - Centrum Medyczne AMED, Lodz
  - Zespol Poradni Specjalistycznych REUMED, Lublin
  - SOLUMED Centrum Medyczne, Poznan
  - Centrum Badan Klinicznych S.C., Poznan
  - Ai Centrum Medyczne Sp. Z O.O. Sp.K., Poznan
  - RCMed, Sochaczew
  - Medycyna Kliniczna, Warsaw
  - Centrum Medyczne AMED, Warsaw
- Clinica GAIAS, Santiago, Spain
- Ukraine (21):
  - CI Dnipropetrovsk CMCH #4 RC, Dnipro
  - Regional CH Dep of Rheumatology SHEI Ivano-Frankivsk NMU, Ivano-Frankivsk
  - GI L.T.Malaya Therapy National Institute of the NAMS of Ukraine, Kharkiv
  - CHI Kharkiv City Clinical Hospital #13, Kharkiv
  - CI A.and O. Tropiny City Clinical Hospital, Kherson
  - Medical Center of Limited Liability Company Medical Clinic Blagomed, Kyiv
  - Med Center 'Ok!Clinic+' of International Institute of Clinical Trials LLC, Kyiv
  - SI NSС M.D. Strazhesko Institute of Cardiology of NAMSU, Kyiv
  - Limited Liability Company Medical Center Concilium Medical, Kyiv
  - LLC Treatment-Diagnostic Center ADONIS plus, Kyiv
  - Volyn Regional Clinical Hospital, Lutsk
  - Lviv Regional Clinical Hospital Dept of Rheumatology NMU, Lviv
  - Mil&Med Cl C of Lviv of the St Border Service of Ukraine, Lviv
  - Center of Reconstructive & Restorative Medicine of Odessa National Medical University, Odesa
  - M.V. Sklifosovskyi Poltava RCH Dept of Rheumatology HSEIU UMSA, Poltava
  - Ternopil University Hospital, Dept. of Rheumatology, SHEI I.Ya.Horbachevskyi Ternopil SMU, Ternopil
  - Private Small Enterprise Medical Center Pulse, Vinnytsia
  - Vinnytsia M.I.Pyrogov RCH Dept of cardiology NMU, Vinnytsia
  - MCIC Health Clinic BO LTD TDC Slaomed, Vinnytsia
  - CI CCH #6 Dept of Therapy ZSMU, Zaporizhzhya
  - CI Zaporizhzhia Regional Clinical Hospital of ZRC, Zaporizhzhya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reinisch W, Hellstrom W, Dolhain RJEM, Sikka S, Westhovens R, Mehta R, Ritter T, Seidler U, Golovchenko O, Simanenkov V, Garmish O, Jeka S, Moravcova R, Rajendran V, Le Brun FO, Arterburn S, Watkins TR, Besuyen R, Vanderschueren D. Effects of filgotinib on semen parameters and sex hormones in male patients with inflammatory diseases: results from the phase 2, randomised, double-blind, placebo-controlled MANTA and MANTA-RAy studies. Ann Rheum Dis. 2023 Aug;82(8):1049-1058. doi: 10.1136/ard-2023-224017. Epub 2023 May 3. PMID 37137672
- [Derived] Hellstrom WJG, Dolhain RJEM, Ritter TE, Watkins TR, Arterburn SJ, Dekkers G, Gillen A, Tonussi C, Gilles L, Oortwijn A, Van Beneden K, de Vries DE, Sikka SC, Vanderschueren D, Reinisch W. MANTA and MANTA-RAy: Rationale and Design of Trials Evaluating Effects of Filgotinib on Semen Parameters in Patients with Inflammatory Diseases. Adv Ther. 2022 Jul;39(7):3403-3422. doi: 10.1007/s12325-022-02168-4. Epub 2022 May 25. PMID 35614292

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Bulgaria, Czech Republic, Estonia, Georgia, Latvia, Poland, Spain, and Ukraine. The first participant was screened on 28 May 2019. A total of 308 participants were screened of which 109 participants were randomized into the study.
Pre-assignment Details: There were 3 distinct parts to the study:
  1) Double-Blind Treatment Phase (DB Phase; Day 1 through the Week 13 study visit); 2) Extension Phase (EXT Phase; after the Week 13 study visit and up to Week 156); and 3) Monitoring Phase (up to 52 weeks).
Groups:
- Filgonitib: Participants received filgotinib 200 milligrams (mg) tablet, orally, once daily up to Week 13 in the DB phase. At Week 13, participants who were arthritis responders, were unblinded and received open-label (OL) treatment filgotinib 200 mg, tablet, orally, once daily up to approximately 143 weeks (until Week 156) in the EXT phase and participants who were arthritis nonresponders discontinued blinded study drug and started standard of care (SOC) treatment in the EXT phase. Participants on DB treatment or OL filgotinib who entered the monitoring phase (if their sperm parameters met ≥50% decrease threshold in pre-specified semen parameters) discontinued the study drug and started SOC for up to 52 weeks.
Period: DB Treatment Phase (Through Week 13)
Arm/Group | Filgonitib | Placebo
Started | 54 | 55
Completed | 54 | 53
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2
Period: EXT Phase (Through Week 156)
Arm/Group | Filgonitib | Placebo
Started | 46 (39 arthritis responder participants entered the EXT phase and received OL treatment filgotinib. 7 arthritis nonresponder participants entered the EXT phase and received SOC treatment.) | 49 (26 arthritis responder participants and 23 arthritis nonresponder participants entered the EXT phase and received SOC treatment.)
Completed | 24 | 26
Not Completed | 22 | 23
Not completed — Adverse Event | 5 | 1
Not completed — Pre-Specified Decrease In Sperm Parameters | 16 | 17
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Physician Decision | 0 | 2
Period: Monitoring Phase (52 Weeks)
Arm/Group | Filgonitib | Placebo
Started (At any visit, participants who had a ≥50% decrease in sperm concentration, and/or sperm motility, and/or sperm morphology compared with baseline entered the Monitoring Phase for evaluation of reversibility.) | 27 | 21
Completed | 27 | 20
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all randomized participants who took ≥ 1 dose of double-blind study drug.
Groups:
- Filgonitib: Participants received filgotinib 200 mg tablet, orally, once daily up to Week 13 in the DB phase. At Week 13, participants who were arthritis responders, were unblinded and received OL treatment filgotinib 200 mg, tablet, orally, once daily up to approximately 143 weeks (until Week 156) in the EXT phase and participants who were arthritis nonresponders discontinued blinded study drug and started SOC treatment in the EXT phase. Participants on DB treatment or OL filgotinib who entered the monitoring phase (if their sperm parameters met ≥50% decrease threshold in pre-specified semen parameters) discontinued the study drug and started SOC for up to 52 weeks.
- Total: Total of all reporting groups
Arm/Group | Filgonitib | Placebo | Total
Number analyzed (Participants) | 54 | 55 | 109
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (8.5) | 39 (7.8) | 40 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 54 | 55 | 109
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 53 | 55 | 108
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 54 | 55 | 109
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Sperm Concentration [Mean (Standard Deviation); unit: million sperms/milliliter (mL)] | 71.2 (41.00) | 66.9 (38.72) | 69.0 (39.74)
Total Sperm Count [Mean (Standard Deviation); unit: million sperms/ejaculate] | 208.4 (136.94) | 225.2 (137.39) | 216.9 (136.79)
Sperm Total Motility [Mean (Standard Deviation); unit: percentage of motile sperm] | 55.9 (8.99) | 58.2 (8.48) | 57.1 (8.77)
Ejaculate Volume [Mean (Standard Deviation); unit: mL] | 3.1 (1.26) | 3.5 (1.29) | 3.3 (1.29)
Percent Normal Sperm Morphology [Mean (Standard Deviation); unit: percentage of normal sperm] | 43 (6.2) | 43 (6.0) | 43 (6.0)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a ≥ 50% Decrease From Baseline in Sperm Concentration at Week 13
Description: Baseline for sperm/semen parameters was the mean of 2 evaluable semen samples at screening. The normal range for sperm concentration is ≥15 million sperms/mL.
  Percentage change = ([mean at Week 13 - baseline] / baseline) × 100; value at Week 13 was the mean of 2 evaluable samples collected at Week 13.
Time Frame: Baseline to Week 13
Population: The Semen Analysis Set included all randomized and treated (≥ 1 dose of double-blind study drug) participants who had 2 semen samples that were eligible for mean calculation at baseline and at the Week 13 analysis visit with the date of the first chronologic semen sample used for purposes of assigning analysis visit windows.
Measure: Number; unit: percentage of participants
Arm/Group | Filgonitib | Placebo
Number analyzed (Participants) | 54 | 53
percentage of participants | 13.0 | 7.5
Statistical Analysis 1: Comparison: Filgonitib vs Placebo; Test type: Other; Difference in Percentage = 5.8, 95% CI 2-sided [-7.5 to 19.2] — Difference in percentage and 95% confidence interval (CI) was based on a stratified Mantel-Haenszel test

2. Secondary Outcome: Percentage of Participants With a ≥ 50% Decrease From Baseline in Sperm Concentration at Week 26
Description: Arthritis responder: For rheumatoid arthritis (RA), psoriatic arthritis (PsA), ankylosing spondylitis (AS), and non-radiographic axial spondyloarthritis (nrAxSpA), a participant with an improvement in the Physician's Global Assessment of Disease Activity (PhGADA) of at least 20% compared with baseline (Day 1) at the specified assessment time.
  Arthritis nonresponder: For RA, PsA, AS, or nrAxSpA, a participant who did not fulfill the definition of arthritis responder at the specified assessment timepoint.
  PhGADA: Physician measured the participant's disease severity on a visual analogue scale (VAS) ranged from 0 (no disease)-100 (worst disease) millimeters (mm).
  Baseline value for sperm/semen parameters was the mean of 2 evaluable semen collections at the screening visit. The normal range for sperm concentration is ≥15 million sperms/mL.
  Percentage change = ([mean at Week 26 - baseline] / baseline) × 100; value at Week 26 was the mean of 2 evaluable samples collected at Week 26.
Time Frame: Baseline to Week 26
Population: The Week 26 Semen Analysis Set included all participants treated (≥ 1 dose of open-label filgotinib or SOC in the extension phase) who had 2 evaluable samples at baseline and at Week 26.
Measure: Number; unit: percentage of participants
Groups:
- Filgotinib/OL Filgotinib (Responder): Participants received filgotinib 200 mg tablet, orally, once daily up to Week 13 in the DB phase. At Week 13, participants who were arthritis responders, were unblinded and received OL treatment filgotinib 200 mg, tablet, orally, once daily up to approximately 143 weeks (until Week 156) in the EXT phase.
- Placebo/SOC (Responder): Participants received placebo (matched to filgotinib) tablet, orally, once daily up to Week 13 in the DB phase. At Week 13, participants who were arthritis responders, were unblinded and started SOC treatment in the EXT phase for up to approximately 143 weeks (until Week 156).
- Filgotinib/SOC (Nonresponder): Participants received filgotinib 200 mg tablet, orally, once daily up to Week 13 in the DB phase. At Week 13, participants who were arthritis nonresponders discontinued blinded study drug and started SOC treatment in the EXT phase for up to approximately 143 weeks (until Week 156).
- Placebo/SOC (Nonresponder): Participants received placebo (matched to filgotinib) tablet, orally, once daily up to Week 13 in the DB phase. At Week 13, participants who were arthritis nonresponders, were unblinded and started SOC treatment in the EXT phase for up to approximately 143 weeks (until Week 156).
Arm/Group | Filgotinib/OL Filgotinib (Responder) | Placebo/SOC (Responder) | Filgotinib/SOC (Nonresponder) | Placebo/SOC (Nonresponder)
Number analyzed (Participants) | 39 | 25 | 7 | 23
percentage of participants | 10.3 | 8.0 | 14.3 | 0

3. Secondary Outcome: Change From Baseline in Sperm Total Motility at Week 13
Description: The normal range for sperm total motility is ≥40%.
Time Frame: Baseline, Week 13
Population: Participants in the Semen Analysis Set with available data were analyzed.
Measure: Median (95% Confidence Interval); unit: percentage of motile sperms
Arm/Group | Filgonitib | Placebo
Number analyzed (Participants) | 54 | 52
percentage of motile sperms | -2.3 [-8.1 to 1.4] | -1.7 [-5.8 to 0.7]
Statistical Analysis 1: Comparison: Filgonitib vs Placebo; Test type: Other; Median Difference (Final Values) = -1.5, 95% CI 2-sided [-6.4 to 3.5] — Difference in Medians and 95% CI for change from baseline at Week 13 was based on quantile regression

4. Secondary Outcome: Change From Baseline in Sperm Total Motility at Week 26
Description: Arthritis responder: For RA, PsA, AS, and nrAxSpA, a participant with an improvement in the PhGADA of at least 20% compared with baseline (Day 1) at the specified assessment time.
  Arthritis nonresponder: For RA, PsA, AS, or nrAxSpA, a participant who did not fulfill the definition of arthritis responder at the specified assessment timepoint.
  PhGADA: Physician measured the participant's disease severity on a VAS ranged from 0 (no disease)-100 (worst disease) mm.
  The normal range for sperm total motility is ≥40%.
Time Frame: Baseline, Week 26
Population: Participants in the Week 26 Semen Analysis Set with available data were analyzed.
Measure: Median (95% Confidence Interval); unit: percentage of motile sperms
Arm/Group | Filgotinib/OL Filgotinib (Responder) | Placebo/SOC (Responder) | Filgotinib/SOC (Nonresponder) | Placebo/SOC (Nonresponder)
Number analyzed (Participants) | 38 | 25 | 7 | 23
percentage of motile sperms | -2.4 [-9.3 to 1.0] | 0.9 [-5.2 to 6.3] | -1.4 [-13.3 to 13.0] | -2.8 [-8.5 to 2.9]

5. Secondary Outcome: Change From Baseline in Total Sperm Count at Week 13
Description: The normal range for total sperm count is ≥ 39 million sperms/ejaculate.
Time Frame: Baseline, Week 13
Population: Participants in the Semen Analysis Set were analyzed.
Measure: Median (95% Confidence Interval); unit: million sperms/ejaculate
Arm/Group | Filgonitib | Placebo
Number analyzed (Participants) | 54 | 53
million sperms/ejaculate | -2.1 [-41.7 to 31.0] | -9.6 [-36.2 to 18.0]
Statistical Analysis 1: Comparison: Filgonitib vs Placebo; Test type: Other; Median Difference (Final Values) = -0.2, 95% CI 2-sided [-37.1 to 36.8] — Difference in medians and 95% CI for change from baseline at Week 13 was based on quantile regression

6. Secondary Outcome: Change From Baseline in Total Sperm Count at Week 26
Description: Arthritis responder: For RA, PsA, AS, and nrAxSpA, a participant with an improvement in the PhGADA of at least 20% compared with baseline (Day 1) at the specified assessment time.
  Arthritis nonresponder: For RA, PsA, AS, or nrAxSpA, a participant who did not fulfill the definition of arthritis responder at the specified assessment timepoint.
  PhGADA: Physician measured the participant's disease severity on a VAS ranged from 0 (no disease)-100 (worst disease) mm.
  The normal range for total sperm count is ≥ 39 million sperms/ejaculate.
Time Frame: Baseline, Week 26
Population: Participants in the Week 26 Semen Analysis Set were analyzed.
Measure: Median (95% Confidence Interval); unit: million sperms/ejaculate
Arm/Group | Filgotinib/OL Filgotinib (Responder) | Placebo/SOC (Responder) | Filgotinib/SOC (Nonresponder) | Placebo/SOC (Nonresponder)
Number analyzed (Participants) | 39 | 25 | 7 | 23
million sperms/ejaculate | -0.2 [-39.5 to 44.5] | 16.8 [-49.3 to 60.6] | 32.2 [-60.8 to 121.3] | -29.9 [-79.8 to 36.6]

7. Secondary Outcome: Change From Baseline in Sperm Concentration at Week 13
Description: The normal range for sperm concentration is ≥15 million sperms/mL.
Time Frame: Baseline, Week 13
Population: Participants in the Semen Analysis Set were analyzed.
Measure: Median (95% Confidence Interval); unit: million sperms/mL
Arm/Group | Filgonitib | Placebo
Number analyzed (Participants) | 54 | 53
million sperms/mL | 3.7 [-7.2 to 13.1] | -0.4 [-6.1 to 7.8]
Statistical Analysis 1: Comparison: Filgonitib vs Placebo; Test type: Other; Median Difference (Final Values) = 7.4, 95% CI 2-sided [-6.0 to 20.8] — Difference in Medians and 95% CI for change from baseline at Week 13 was based on quantile regression

8. Secondary Outcome: Change From Baseline in Sperm Concentration at Week 26
Description: Arthritis responder: For RA, PsA, AS, and nrAxSpA, a participant with an improvement in the PhGADA of at least 20% compared with baseline (Day 1) at the specified assessment time.
  Arthritis nonresponder: For RA, PsA, AS, or nrAxSpA, a participant who did not fulfill the definition of arthritis responder at the specified assessment timepoint.
  PhGADA: Physician measured the participant's disease severity on a VAS ranged from 0 (no disease)-100 (worst disease) mm.
  The normal range for sperm concentration is ≥15 million sperms/mL.
Time Frame: Baseline, Week 26
Population: Participants in the Week 26 Semen Analysis Set were analyzed.
Measure: Median (95% Confidence Interval); unit: million sperms/mL
Arm/Group | Filgotinib/OL Filgotinib (Responder) | Placebo/SOC (Responder) | Filgotinib/SOC (Nonresponder) | Placebo/SOC (Nonresponder)
Number analyzed (Participants) | 39 | 25 | 7 | 23
million sperms/mL | 1.7 [-8.9 to 21.2] | 9.6 [-3.7 to 29.0] | 10.3 [-43.5 to 36.3] | -5.8 [-12.9 to 4.6]

9. Secondary Outcome: Change From Baseline in Ejaculate Volume at Week 13
Description: The normal range for ejaculate volume is ≥1.5 mL.
Time Frame: Baseline, Week 13
Population: Participants in the Semen Analysis Set were analyzed.
Measure: Median (95% Confidence Interval); unit: mL
Arm/Group | Filgonitib | Placebo
Number analyzed (Participants) | 54 | 53
mL | -0.3 [-0.6 to 0.1] | -0.2 [-0.4 to 0.1]
Statistical Analysis 1: Comparison: Filgonitib vs Placebo; Test type: Other; Median Difference (Final Values) = -0.3, 95% CI 2-sided [-0.6 to 0.1] — Difference in Medians and 95% CI for change from baseline at Week 13 was based on quantile regression

10. Secondary Outcome: Change From Baseline in Ejaculate Volume at Week 26
Description: Arthritis responder: For RA, PsA, AS, and nrAxSpA, a participant with an improvement in the PhGADA of at least 20% compared with baseline (Day 1) at the specified assessment time.
  Arthritis nonresponder: For RA, PsA, AS, or nrAxSpA, a participant who did not fulfill the definition of arthritis responder at the specified assessment timepoint.
  PhGADA: Physician measured the participant's disease severity on a VAS ranged from 0 (no disease)-100 (worst disease) mm.
  The normal range for ejaculate volume is ≥1.5 mL.
Time Frame: Baseline, Week 26
Population: Participants in the Week 26 Semen Analysis Set were analyzed.
Measure: Median (95% Confidence Interval); unit: mL
Arm/Group | Filgotinib/OL Filgotinib (Responder) | Placebo/SOC (Responder) | Filgotinib/SOC (Nonresponder) | Placebo/SOC (Nonresponder)
Number analyzed (Participants) | 39 | 25 | 7 | 23
mL | -0.2 [-0.7 to 0.4] | -0.6 [-0.7 to -0.2] | 0.2 [-1.0 to 1.1] | -0.3 [-0.6 to 0.2]

11. Secondary Outcome: Change From Baseline in Percent Normal Sperm Morphology at Week 13
Description: The normal range for percent normal sperm morphology is ≥30% normal sperms.
Time Frame: Baseline, Week 13
Population: Participants in the Semen Analysis Set were analyzed.
Measure: Median (95% Confidence Interval); unit: percentage of normal sperms
Arm/Group | Filgonitib | Placebo
Number analyzed (Participants) | 54 | 53
percentage of normal sperms | 1 [-1 to 2] | 1 [-1 to 3]
Statistical Analysis 1: Comparison: Filgonitib vs Placebo; Test type: Other; Median Difference (Final Values) = -1, 95% CI 2-sided [-3 to 1] — Difference in Medians and 95% CI for change from baseline at Week 13 was based on quantile regression

12. Secondary Outcome: Change From Baseline in Percent Normal Sperm Morphology at Week 26
Description: Arthritis responder: For RA, PsA, AS, and nrAxSpA, a participant with an improvement in the PhGADA of at least 20% compared with baseline (Day 1) at the specified assessment time.
  Arthritis nonresponder: For RA, PsA, AS, or nrAxSpA, a participant who did not fulfill the definition of arthritis responder at the specified assessment timepoint.
  PhGADA: Physician measured the participant's disease severity on a VAS ranged from 0 (no disease)-100 (worst disease) mm.
  The normal range for percent normal sperm morphology is ≥30% normal sperms.
Time Frame: Baseline, Week 26
Population: Participants in the Week 26 Semen Analysis Set were analyzed.
Measure: Median (95% Confidence Interval); unit: percentage of normal sperms
Arm/Group | Filgotinib/OL Filgotinib (Responder) | Placebo/SOC (Responder) | Filgotinib/SOC (Nonresponder) | Placebo/SOC (Nonresponder)
Number analyzed (Participants) | 39 | 25 | 7 | 23
percentage of normal sperms | 1 [-2 to 5] | 3 [-2 to 8] | 3 [-15 to 6] | 4 [1 to 8]

ADVERSE EVENTS:
Time Frame: From first dose up to Week 156. TEAEs were considered as AEs with onset on or after the first dose of study drug to the last dose + 30 days. AEs leading to premature discontinuation study drug was also a TEAE.
Description: The Safety Analysis Set included all randomized participants who took ≥ 1 dose of double-blind study drug. The Extension Phase Safety Analysis Set included all participants who took ≥ 1 dose of open-label filgotinib or standard of care in the extension phase of the study.
Groups:
- Double-Blind Phase: Filgotinib 200 mg: Participants received filgotinib 200 mg tablet, orally, once daily up to Week 13 in the DB phase.
- Double-Blind Phase: Placebo: Participants received placebo (matched to filgotinib) tablet, orally, once daily up to Week 13 in the DB phase.
- Extension Phase: Placebo - SOC: At Week 13, participants were unblinded and started SOC treatment in the EXT phase, for up to approximately 143 weeks (until Week 156).
- Extension Phase: Filgotinib 200 mg - SOC: At Week 13, participants who were arthritis nonresponders discontinued blinded study drug and started SOC treatment in the EXT phase, for up to approximately 143 weeks (until Week 156).
- Extension Phase: Filgotinib 200 mg - OL Filgotinib 200 mg: At Week 13, participants who were arthritis responders, were unblinded and received OL treatment filgotinib 200 mg, tablet, orally, once daily in the EXT phase, for up to approximately 143 weeks (until Week 156).
Arm/Group | Double-Blind Phase: Filgotinib 200 mg | Double-Blind Phase: Placebo | Extension Phase: Placebo - SOC | Extension Phase: Filgotinib 200 mg - SOC | Extension Phase: Filgotinib 200 mg - OL Filgotinib 200 mg
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/55 | 0/49 | 0/7 | 0/39
Serious Adverse Events (participants affected / at risk) | 2/54 | 1/55 | 2/49 | 1/7 | 5/39
Other Adverse Events (participants affected / at risk) | 12/54 | 10/55 | 23/49 | 5/7 | 20/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-Blind Phase: Filgotinib 200 mg (N=54) | Double-Blind Phase: Placebo (N=55) | Extension Phase: Placebo - SOC (N=49) | Extension Phase: Filgotinib 200 mg - SOC (N=7) | Extension Phase: Filgotinib 200 mg - OL Filgotinib 200 mg (N=39)
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Uveitis (Eye disorders) | 0 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double-Blind Phase: Filgotinib 200 mg (N=54) | Double-Blind Phase: Placebo (N=55) | Extension Phase: Placebo - SOC (N=49) | Extension Phase: Filgotinib 200 mg - SOC (N=7) | Extension Phase: Filgotinib 200 mg - OL Filgotinib 200 mg (N=39)
Hypertension (Vascular disorders) | 2 | 2 | 1 | 0 | 2
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 1 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 2 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 2 | 0 | 2
Headache (Nervous system disorders) | 2 | 1 | 2 | 1 | 2
Sciatica (Nervous system disorders) | 0 | 0 | 1 | 1 | 0
External ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 2
Splenic artery aneurysm (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Renal aneurysm (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 10 | 3 | 6
Herpes zoster disseminated (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Latent tuberculosis (Infections and infestations) | 0 | 0 | 1 | 0 | 3
Nasopharyngitis (Infections and infestations) | 4 | 4 | 3 | 4 | 2
Pharyngitis (Infections and infestations) | 2 | 2 | 2 | 0 | 2
Pyospermia (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 3 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 3 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 3 | 0 | 2
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 1 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 2
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must review and approve any results of the study or abstracts for professional meetings prepared by the investigator(s). Published data must not compromise the objectives of the study. Data from individual study centers in multicenter studies must not be published separately.

DOCUMENTS (2):
  • Study Protocol (2022-09-09): https://cdn.clinicaltrials.gov/large-docs/95/NCT03926195/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-12): https://cdn.clinicaltrials.gov/large-docs/95/NCT03926195/SAP_001.pdf